CLINICAL TRIAL: NCT02223364
Title: Prospective, Randomized, Controlled Trial Comparing Continuous Femoral and Single Injection Sciatic Peripheral Nerve Blocks vs Periarticular Injection With Ropivacaine or Liposomal Bupivacaine (Exparel) on Patients Undergoing Total Knee Arthroplasty
Brief Title: Peripheral Nerve Blocks vs Periarticular Local Anesthetic Injection for Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sandra (Sandy) L. Kopp, M.D., Associate Professor of Anesthesiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-002083
Record Dates: First submitted 2014-07-29; First posted 2014-08-22 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Bupivacaine; Injections, Intra-Articular; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Peripheral Nerve Block (PNB) (Active Comparator): This group received a continuous femoral nerve block and a single injection sciatic nerve block consisting of the following: Peripheral nerve blocks with Bupivacaine.
  Interventions: Drug: Peripheral nerve blocks with Bupivacaine
- Ropivacaine (PAI-R) (Active Comparator): This group received intra articular injection with Ropivacaine, a total volume of 120 milliliters (mL) injected in the periarticular structures by the surgeon. Following the current, standardized practice for periarticular infiltration, approximately 30 - 40 mL of solution was injected into the posterior capsule just prior to cementing the implants in place and 40 - 50 mL of solution injected into the medial and lateral retinaculum while the cement was hardening and prior to deflation of the tourniquet. The remaining volume of approximately 40 mL was injected into the quadriceps tendon and subcutaneous tissue prior to skin closure.
  Interventions: Drug: Intra articular injection with Ropivacaine
- Liposomal Bupivacaine (PAI-L) (Active Comparator): This group received Intra articular injection with liposomal bupivacaine, a total volume of 120 milliliters (mL) injected in the periarticular structures by the surgeon. Following the current, standardized practice for periarticular infiltration, approximately 30 - 40 mL of solution was injected into the posterior capsule just prior to cementing the implants in place and 40 - 50 mL of solution injected into the medial and lateral retinaculum while the cement was hardening and prior to deflation of the tourniquet. The remaining volume of approximately 40 mL was injected into the quadriceps tendon and subcutaneous tissue prior to skin closure.
  Interventions: Drug: Intra articular injection with liposomal bupivacaine

INTERVENTIONS:
Drug: Peripheral nerve blocks with Bupivacaine — Subjects received Bupivacaine 0.5% preoperatively, then Bupivacaine 0.2% upon post anesthesia care unit (PACU) arrival via femoral nerve block, then Bupivacaine 0.25% via single-injection sciatic nerve.
  Other Names: Marcaine; Sensorcaine
  Arms: Peripheral Nerve Block (PNB)
Drug: Intra articular injection with Ropivacaine — Subjects received an intra articular injection with Ropivacaine, a total volume of 120 milliliters (mL) injected in the periarticular structures by the surgeon. Ropivacaine dose depended upon body weight: 50-74.9 kg: 200 mg, 75-99.9 kg: 300 mg, 100-125 kg: 400 mg.
  Other Names: Naropin
  Arms: Ropivacaine (PAI-R)
Drug: Intra articular injection with liposomal bupivacaine — Subjects received an intra articular injection with liposomal bupivacaine, a total volume of 120 mL injected in the periarticular structures by the surgeon. Patients weighing 50-125 kg received 266mg of Liposomal Bupivacaine.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine (PAI-L)

SUMMARY:
The purpose of this study is to find a better way to make patients comfortable after their knee surgery. The investigators compared three ways of providing pain relief, either by use of a nerve block at the femoral and sciatic nerve areas, or with actual injections in the surgical joint area with one of two different medicines, either ropivacaine or liposomal bupivacaine (Exparel®). The hypothesis was that the nerve block at the femoral and sciatic nerve areas would result in lower pain scores and opioid consumption than either of the two injections in the surgical joint area.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with an American Society of Anesthesiologists (ASA) physiological status I-III
2. Patients presenting for unilateral primary total knee replacement.
3. No focal neurologic deficit of the surgical lower extremity.
4. Cognitively intact with the ability to sign informed consent

Exclusion Criteria:

1. Chronic pain syndromes such as fibromyalgia or complex regional pain syndrome
2. History of long term use of daily opioids (>1 months) with oral morphine equivalent (OME) >5mg/day.
3. Body mass index (BMI) > 40 kg/m2
4. Allergies to medications used in this study such as: fentanyl, hydromorphone, ketorolac, ibuprofen, acetaminophen, local anesthetics, oxycodone, OxyContin, tramadol, ondansetron, droperidol, or dexamethasone, celecoxib
5. Major systemic medical problems such as:

   * Severe renal disorder defined as glomerular filtration rate (GFR) <50 units/m2
   * Cardiovascular disorders defined as congestive heart failure (CHF) New York Heart Association (NYHA) class III-IV
   * Severe hepatic disorder defined as current or past diagnosis of acute/subacute necrosis liver, acute hepatic failure, chronic liver disease, cirrhosis (primary biliary cirrhosis), fatty liver, chronic hepatitis/toxic hepatitis, liver abscess, hepatic coma, hepatorenal syndrome, other disorders of liver.
6. Impaired cognitive function or inability to understand the study protocol
7. Contraindication to a regional anesthesia technique (e.g., preexisting neuropathy in the operative extremity, coagulopathy [platelets < 100,000, International Normalized Ratio (INR) >1.5], refusal, etc.).
8. Previous contralateral knee replacement managed with regional or periarticular injection
9. Unable to follow-up at the 3 month interval at Mayo Clinic in Rochester, Minnesota
10. Pregnancy or breast feeding (women of child-bearing potential, must have a negative pregnancy test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Kopp, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amundson AW, Johnson RL, Abdel MP, Mantilla CB, Panchamia JK, Taunton MJ, Kralovec ME, Hebl JR, Schroeder DR, Pagnano MW, Kopp SL. A Three-arm Randomized Clinical Trial Comparing Continuous Femoral Plus Single-injection Sciatic Peripheral Nerve Blocks versus Periarticular Injection with Ropivacaine or Liposomal Bupivacaine for Patients Undergoing Total Knee Arthroplasty. Anesthesiology. 2017 Jun;126(6):1139-1150. doi: 10.1097/ALN.0000000000001586. PMID 28234636

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Mayo Clinic in Rochester, Minnesota from October 2014 to December 2015.
Period: Overall Study
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Started | 55 | 55 | 55
Completed | 50 | 55 | 52
Not Completed | 5 | 0 | 3
Not completed — Protocol Violation | 3 | 0 | 3
Not completed — subject expired before surgery | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L) | Total
Number analyzed (Participants) | 50 | 55 | 52 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9) | 68 (8) | 67 (8) | 67.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 34 | 27 | 86
  Male | 25 | 21 | 25 | 71
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 55 | 52 | 157

OUTCOME MEASURES:

1. Primary Outcome: Maximum Pain Post-Operative Day (POD) 1 (Morning)
Description: Pain was measured on a 1-10 numeric pain rating scale (NRS) with 0=no pain, and 10=worst pain imaginable.
Time Frame: Post-Operative Day 1, approximately 6 am to 12:00 pm
Population: Intent-to-Treat Analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
units on a scale | 3 [1 to 6] | 4 [2 to 6] | 4.5 [3 to 6]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.144, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.196, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Average Pain Post-Postanesthesia Care Unit (PACU)
Description: Pain was measured on a 1-10 numeric pain rating scale (NRS) with 0=no pain, and 10=worst pain imaginable.
Time Frame: Post-operative Day 0, approximately 12 pm to 12 am
Population: Intent-to-Treat analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
units on a scale | 0.6 [0.0 to 2.2] | 1.7 [0.9 to 2.5] | 2.4 [1.1 to 3.6]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Maximum Pain Post-PACU
Description: Pain was measured on a 1-10 numeric pain rating scale (NRS) with 0=no pain, and 10=worst pain imaginable.
Time Frame: Post-operative Day 0, approximately 12 pm to 12 am
Population: Intent-to-Treat Analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
units on a scale | 1 [0 to 4] | 4 [2 to 6] | 5 [3 to 6]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.257, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Average Pain POD 1 (24 Hours)
Description: Pain was measured on a 1-10 numeric pain rating scale (NRS) with 0=no pain, and 10=worst pain imaginable.
Time Frame: POD 1, approximately 12 am to 12 am next day
Population: Intent-to-Treat Analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
units on a scale | 2.5 [1.2 to 4.2] | 3.5 [2.5 to 4.6] | 3.7 [2.9 to 4.6]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.059, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.214, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Maximum Pain POD 1 (24 Hours)
Description: Pain was measured on a 1-10 numeric pain rating scale (NRS) with 0=no pain, and 10=worst pain imaginable.
Time Frame: POD 1, approximately 12 am to 12 am next day
Population: Intent-to-Treat Analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
units on a scale | 5.5 [3 to 7] | 6 [5 to 7] | 6 [5 to 8]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.189, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.043, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.357, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Average Pain POD 2 (24 Hours)
Description: Pain was measured on a 1-10 numeric pain rating scale (NRS) with 0=no pain, and 10=worst pain imaginable.
Time Frame: POD 2, approximately 12 am to 12 am next day
Population: Intent-to-Treat Analysis. For POD 2, data are missing for 5 subjects (1 on Peripheral Nerve Block (PNB) arm, 1 on Ropivacaine (PAI-R) arm, and 3 on Liposomal Bupivacaine (PAI-L) arm).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 49 | 54 | 49
units on a scale | 3.3 [2.0 to 4.2] | 3.2 [2.4 to 4.0] | 3.5 [2.8 to 4.3]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.958, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.203, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.132, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Maximum Pain POD 2 (24 Hours)
Description: Pain was measured on a 1-10 numeric pain rating scale (NRS) with 0=no pain, and 10=worst pain imaginable.
Time Frame: POD 2, approximately 12 am to 12 am next day
Population: Intent-to-Treat Analysis. For POD 2, data are missing for 5 subjects (1 on PNB arm, 1 on PAI-R arm, and 3 on PAI-L arm).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 49 | 54 | 49
units on a scale | 5 [3 to 7] | 6 [4 to 7] | 6 [5 to 7]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.493, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.299, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.797, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Preoperative Daily Opioid Use
Description: Opioid consumption will be documented in the patient electronic medical record by the nursing staff caring for the patient.
Time Frame: baseline
Population: Intent-to-Treat Analysis
Measure: Median (Inter-Quartile Range); unit: mg oral morphine equivalents (OME)
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
mg oral morphine equivalents (OME) | 15 [0 to 15] | 15 [0 to 15] | 15 [1 to 15]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.571, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.991, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.496, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Intraoperative Opioid Use
Description: Opioid consumption was documented in the patient electronic medical record by the nursing staff caring for the patient.
Time Frame: During the procedure, approximately 2 hours after start of the procedure
Population: Intent-to-treat analysis
Measure: Median (Inter-Quartile Range); unit: mg OME
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
mg OME | 10 [5 to 15] | 10 [5 to 15] | 10 [7 to 20]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.807, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.171, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R); Test type: Superiority; p = 0.104, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: PACU Opioid Use
Description: Opioid consumption was documented in the patient electronic medical record by the nursing staff caring for the patient.
Time Frame: Approximately 2 hours after entry in PACU
Population: Intent-to-treat analysis
Measure: Median (Inter-Quartile Range); unit: mg OME
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
mg OME | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

11. Secondary Outcome: POD 0 Post-PACU Opioid Use
Description: Additional opioid medications that were taken by subjects (recorded at the same time as the time points for measuring pain). Opioid consumption was documented in the patient electronic medical record by the nursing staff caring for the patient.
Time Frame: POD 0, approximately 12 pm to 12 am
Population: Intent-to-treat
Measure: Median (Inter-Quartile Range); unit: mg OME
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
mg OME | 0 [0 to 15] | 8 [0 to 30] | 15 [0 to 30]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.293, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: POD 1 Opioid Use
Description: as for outcome 11
Time Frame: POD 1, approximately 12 am to 12 am next day
Population: Intent-to-treat analysis
Measure: Median (Inter-Quartile Range); unit: mg OME
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
mg OME | 26 [0 to 53] | 38 [15 to 53] | 45 [15 to 82]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.202, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.148, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: POD 2 Opioid Use
Description: as for outcome 11
Time Frame: POD 2, approximately 12 am to 12 am next day
Population: Intent-to-treat analysis. For POD 2, data are missing for 5 subjects (1 on PNB arm, 1 on PAI-R arm, and 3 on PAI-L arm).
Measure: Median (Inter-Quartile Range); unit: mg OME
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 49 | 54 | 49
mg OME | 23 [0 to 38] | 15 [0 to 38] | 23 [15 to 45]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R); Test type: Superiority; p = 0.933, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Peripheral Nerve Block (PNB) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.169, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.126, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Hospital Length of Stay
Description: The hospital length of stay was measured from the date of admittance until the date of discharge.
Time Frame: Approximately 3 days
Population: Intent-to-treat analysis
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
days | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB) vs Ropivacaine (PAI-R) vs Liposomal Bupivacaine (PAI-L); Test type: Superiority; p = 0.768, Kruskal-Wallis

15. Secondary Outcome: Balance Testing on Operative Leg Using Unipedal Stance Time
Description: In order to measure clinical balance, unipedal stance time (UST) was collected as an indicator of balance and fall risk. Timing (in seconds) began upon withdrawal of support and continued until the uplifted foot returned to the floor, the subject required support, or if the subject reached a time limit of 30 seconds. The best performance of three repetitions was recorded for analysis. Normative values for the UST are available. A UST threshold of 30 seconds yields a sensitivity of 95% and a specificity of 58% in identifying those with a history of falls. The first five seconds of unipedal stance is indicative of dynamic balance; inability to maintain unipedal stance for five seconds is a significant predictor of injurious falls.
Time Frame: baseline, approximately 12 weeks
Population: Intent-to-treat analysis
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
Number analyzed (Participants) | 50 | 55 | 52
seconds
  baseline | 24 [7 to 30] | 16 [5 to 30] | 17 [3 to 30]
  12 weeks | 20 [8 to 30] | 30 [11 to 30] | 23 [8 to 30]
Statistical Analysis 1: Comparison: Peripheral Nerve Block (PNB); Within group comparison of baseline and 3 months (approximately 12 weeks); Test type: Superiority; p = 0.623, Regression, Cox
Statistical Analysis 2: Comparison: Ropivacaine (PAI-R); Within group comparison of baseline and 3 months (approximately 12 weeks); Test type: Superiority; p = 0.001, Regression, Cox
Statistical Analysis 3: Comparison: Liposomal Bupivacaine (PAI-L); Within group comparison of baseline and three months (approximately 12 weeks); Test type: Superiority; p = 0.048, Regression, Cox

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Peripheral Nerve Block (PNB) | Ropivacaine (PAI-R) | Liposomal Bupivacaine (PAI-L)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/55 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/55 | 0/52
Other Adverse Events (participants affected / at risk) | 2/50 | 3/55 | 3/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral Nerve Block (PNB) (N=50) | Ropivacaine (PAI-R) (N=55) | Liposomal Bupivacaine (PAI-L) (N=52)
Fall (General disorders) | 2 (2) | 1 (1) | 1 (1) — 2 in the peripheral nerve block group fell during their hospital stay; one in the ropivacaine periarticular injection group and one in the liposomal bupivacaine periarticular injection group fell after hospital discharge.
Superficial wound infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) — Six patients, two in each group experienced a superficial wound infection after hospital discharge that required treatment with antibiotics.
Rapid Response Team (General disorders) | 0 (0) | 1 (1) | 1 (1) — Adverse event occurred during the patients' hospital stay.
Nerve Injury (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) — This adverse event occurred after hospital discharge.
Additional surgery (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes